CLINICAL TRIAL: NCT01776203
Title: Initiation of Medical Menopause With Depot Leuprolide Acetate vs Depot Leuprolide Acetate Plus Medroxyprogesterone Acetate: A Pilot Randomized
Brief Title: Study of a Progestin to Prevent Bleeding Associated With Initiation of Medical Menopause With GnRH Agonist
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20110523
Record Dates: First submitted 2011-06-14; First posted 2013-01-28 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Dysfunctional Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- medroxyprogesterone acetate (Active Comparator)
  Interventions: Drug: Medroxyprogesterone 17-Acetate
- control (No Intervention)

INTERVENTIONS:
Drug: Medroxyprogesterone 17-Acetate — MPA pills 20 mg (2 X 10 mg) twice daily for 3 weeks
  Other Names: Provera
  Arms: medroxyprogesterone acetate

SUMMARY:
In this study, the investigators would like to see if giving medroxyprogesterone acetate for 3 weeks after Leuprolide acetate injection will help to decrease this amount of bleeding, decrease the amount of nausea, bloating and cramping and increase patient satisfaction

DETAILED DESCRIPTION:
Gonadotrophin releasing hormone is a decapeptide produced in the hypothalamus that stimulates both follicle stimulating hormone and lutenizing hormone secretion from the anterior pituitary in response to a number of endocrine feedback loops that include estradiol, progesterone, and inhibin. Leuprolide acetate is a synthetic decapeptide and a potent gonadrotropin-releasing hormone agonist that can be used in a number of clinical conditions such as endometriosis, chronic pelvic pain, uterine leiomyomas, adenomyosis, central precocious puberty and in-vitro fertilization.

This agonist is more potent that the natural gonadotrophin releasing hormone peptide as it has a stronger affinity for the receptor and also has a longer half-life. Following administration the high levels of gonadrotropin-releasing hormone agonist produce an immediate increase in pituitary luteinizing hormone and follicle stimulating hormone secretion ('flare-up'), which leads to an increase in serum estradiol within 2 days of administration However, unlike the physiological state, where gonadotrophin releasing hormone is produced in a pulsatile fashion, the tonically elevated levels of gonadrotropin-releasing hormone agonist will cause a downregulation of pituitary receptors and desensitization of the pituitary gonadotrophs which leads to a hypogonadotropic state by the fourth week post injection. This suppression is the basis for the clinical application of this drug in gynecology. With the initial 'flare-up', however, there can be an episode of uterovaginal bleeding secondary to the endometrial impact of the temporary, self limited, high circulating levels of estradiol. that appear to in the second week. This bleeding can especially be a cause for concern in women who are already anemic at baseline.

A suggested approach for reducing or preventing this flare-related bleeding is the administration of a progestin or estrogen-progestin combination preparation in conjunction with the initiation of gonadrotropin-releasing hormone agonist therapy. The putative role of the progestin is to reduce the responsiveness of the endometrium to estradiol by downregulating endometrial estrogen receptors. Such an approach could mitigate the impact of the estradiol flare thereby reducing the volume of the flare-related bleeding, or, potentially, eliminate it altogether. However, a systematic review of published literature fails to identify any studies evaluating methods designed to reduce bleeding associated with the gonadrotropin-releasing hormone flare. The databases searched included the Cochrane Database of Systematic Reviews as well MEDLINE using the PubMed search engine. Search words and phrases included: gonadrotropin-releasing hormone agonist, bleeding, gonadrotropin-releasing hormone agonist flare progestin, and leuprolide acetate. The current instructions for use from the FDA for approved gonadrotropin-releasing hormone agonist compounds such as leuprolide acetate do not recommend or mandate the use of progestins with the use of gonadrotropin-releasing hormone agonist. The standard of care at this time, therefore, is that progestins or estrogen-progestin compounds are not used when initiating gonadrotropin-releasing hormone agonist therapy. As a result it seems appropriate to perform structured investigation of the role of progestin-based regimens for the mitigation of gonadrotropin-releasing hormone agonist-induced flare bleeding.

The proposed project is a pilot randomized trial to be performed in selected gonadrotropin-releasing hormone agonist-naieve women who are initiating gonadrotropin-releasing hormone agonist therapy with leuprolide acetate 11.25 mg as determined by their clinicians. The study group will be randomized into one of two arms: Those receiving medroxyprogesterone acetate administered orally in a dose of 20 mg twice daily for the first three weeks after their first leuprolide acetate injection and the "control" group, who receive no progestin therapy. Medroxyprogesterone acetate was selected because it is FDA-approved for abnormal uterine bleeding, it is in widespread use and is well tolerated, and there are multiple studies describing the use of dosages higher than those proposed for this study. One such study was performed and published by our group evaluating daily doses of medroxyprogesterone acetate as high as 60 mg for the treatment of acute uterine bleeding in nongravid patients. If the investigators are able to demonstrate that the use of medroxyprogesterone acetate significantly reduces or eliminates the volume of uterine bleeding associated with the initiation of gonadrotropin-releasing hormone agonist therapy, women in the KP system and elsewhere may be spared this side effect of treatment. Such a finding may have special value for women who are already anemic and, consequently, unable to tolerate a treatment associated bleed.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal women 18-50 years of age
2. Requiring gonadrotropin-releasing hormone agonist for any indication except ovulation induction
3. If there is abnormal uterine bleeding, such bleeding is not obviously related to structural defects such as polyps or submucous leiomyomas; subserosal and intramural myomas (International Federation of Gynecology and Obstetrics Classification 3-8 inclusive) are acceptable

Exclusion Criteria:

1. Currently pregnant
2. Recent used of gonadrotropin-releasing hormone agonist

   1. 1 month depot formulation eg leuprolide acetate 3.75, within 90 days
   2. 3 month depot formulation eg leuprolide acetate 11.25 within 180 days
3. Currently has an intrauterine contraceptive device
4. Currently on gonadal steroids (including birth control pills, rings, or implantable or injectable agents)
5. History of breast cancer
6. Currently undergoing ovulation induction
7. History of adverse reactions to gonadal steroids
8. Hemoglobin <8 mg/dl as measured within 30 days of enrollment (Baseline hemoglobin is standard of care for patients initiating gonadrotropin-releasing hormone agonist therapy)
9. Weight above >250 lbs
10. Has a known submucous leiomyoma ( International Federation of Gynecology and Obstetrics Class type 0, 1, 2)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Amount of bleeding with or without use of medroxyprogesterone acetate after initiation of gonadrotropin-releasing hormone agonist therapy, | 30 days
  The primary outcome of this study will be the amount of bleeding as measured by the validated Mansfield scale experienced by patients in the 28 days following the initiation of GnRHa therapy. This scale is from 0 (no bleeding) to 6 (very heavy bleeding or gushing). The patients will fill out this diary every day for 3 weeks after receiving GnRHa therapy.

SECONDARY OUTCOMES:
the number of days of bleeding, nausea, bloating, and pelvic pain | 30 days
  2.2 Secondary outcomes will include the number of days of bleeding, nausea, bloating, and pelvic pain. These outcomes were set to evaluate efficacy of treatment (amount of bleeding, number of days of bleeding) as well as common side effects experienced with the medications being used (nausea, bloating, pelvic pain). The pelvic pain will be meausured based on a scale from 0 (none) to 10 (worst imaginable pain). Patient's nausea, bloating and breast tenderness is based on a scale from 0 (none) to 4 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Munro, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente, Los Angeles, California, United States